CLINICAL TRIAL: NCT01041300
Title: The Effects of Trancranial Magnetic Stimulation Multichannel Stimulator on Motor Excitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0015-09-SHA
Record Dates: First submitted 2009-12-22; First posted 2009-12-31 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Transcranial Magnetic Stimulation; TMS; Motor Threashold; Multiway; Magstim Rapid 2; Abductor policis brevis; Figure 8 coil; Double cone coil; Circular coil; Brainsway; Healthy participants.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Magstim Rapid2 Stimulator — Duration: Time is takes to find motor thresholds obtained with figure-8 coil using Magstim Rapid2 Stimulator (Estimated at 15 minutes).
  Total Duration of device: 15 minutes
Device: Brainsway Multi-channel Stimulator — Finding motor thresholds using the figure-8 coil and the Brainsway Multi-channel Stimulator (Estimated at 15 minutes).
  Finding motor threshold of leg obtained with Double Cone coil using the Brainsway Multi-channel Stimulator (Estimated at 15 minutes).
  Finding motor threshold of leg obtained with circular coils using the Brainsway Multi-channel Stimulator (Estimated at 15 minutes).
  Finding motor threshold of thumb obtained with circular coils on multiple channels using the Brainsway Multi-channel Stimulator (Estimated at 15 minutes).
  Finding motor thresholds of multiple channels using the Brainsway Multi-channel Stimulator (Estimated at 1 hour).
  Finding specificity of the motor thresholds of multiple channels using the Brainsway Multi-channel Stimulator (Estimated at 30 minutes).
  Total Duration with Device: 2 hours and 30 minutes

SUMMARY:
Our aim is to Test the influence of a new multichanel Transcranial Magnetic Stimulation stimulator (Multiway) on motor excitation, in comparision to a wildly used Magstim Super Rapid 2 single channel stimulator.

Each of the 20 Healthy subjects that are inticipated to inrole to the study wiil undergo 6 simple procedures which are designed to compare the motor threshold obtained by diffrent combination of TMs coils (figure 8, double cone coil,H coil array) and stimulators (Multiway, Super Rapid 2).

The entire length of the procedures is about 4 hours and all subjects will be paid for their participation in the study.

Our main hypothesis is that the motor threshold obtained by the multichanel stimulator will be significtly lower then the single chanel stimulator.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 18-65
2. Right handed individuals
3. Individual provides Negative responses to the questions on the safety questionnaire completed prior to TMS treatment.
4. Individual gave both written and verbal consent to participation in the study.

Exclusion Criteria:

1. Individual suffers from an Axis I disorder, as diagnosed in a Clinical interview with a Psychiatrist.
2. Individual suffers from an Axis II disorder, as diagnosed in a Clinical interview with a Psychiatrist.
3. Individual has a history of high blood pressure.
4. Individual has a history of epilepsy, epileptic seizure, or febrile seizures.
5. Individual has family members with a history of epilepsy, epileptic seizures or febrile seizures.
6. Individual has a history of head injury.
7. Individual has any metal implants in head (except for dental implants)
8. Individual has history of surgery, including metal implants or individual has a known history of metal particals in the eye, heart pumps, neurostimulator use, or any other medical pump.
9. Individual has a history of migrane.
10. Individual has a history of hearing problems or deafness.
11. Individual has a hisotry of hearing aids or implants.
12. Individual has a hisotry of drug or alcohol addiction.
13. Individual is pregnant or is sexually active and not using contraception.
14. Individual is to difficult to contact.
15. Indicidual has a legal gaurdian.
16. Individual is currently enroleld in another medical study.
17. Individual is a soldier, a prisoner or a convict.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Comparison between abductor policis brevis (APB) motor thresholds obtained with figure-8 using Magstim and Brainsway stimulators, for the same subjects | one day
Comparison between the total power required for APB motor thresholds obtained with figure-8 Coil operated with a single channel, and circular coils operated with several channels of the Brainsway stimulator, for the same subjects. | one day
Comparison between the total power required for leg motor thresholds obtained with Double Cone Coil operated with a single channel, and circular coils operated with several channels of the Brainsway stimulator, for the same subjects. | one day
Comparison between the latency times for leg motor thresholds obtained with Double Cone Coil operated with a single channel, and circular coils operated with several channels of the Brainsway stimulator, for the same subjects. | one day
Comparison between the motor thresholds and motor evoked potentials (MEPs) obtained with various combinations of relative intensities of pulses produced by several channels of the multi-channel Brainsway stimulator. | one day

CONTACTS AND LOCATIONS:
Overall Officials: Eiran V Harel, MD, Principal Investigator — Shalvata Mental Health Center
Locations (1):
- Shalvata Mental Health Center, Hod HaSharon, Israel